CLINICAL TRIAL: NCT03996096
Title: Etude Observationnelle Biologique Sur le Syndrome de Sevrage Des Inhibiteurs de Tyrosine Kinase Dans la Leucémie Myéloïde Chronique.
Brief Title: Tyrosine Kinase Inhibitor Withdrawal Syndrome in CML Patients: Observatory Trial Studying the Biological Factors.
Acronym: KIWIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 18-206
Record Dates: First submitted 2019-05-23; First posted 2019-06-24 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-03

CONDITIONS: Chronic Myeloid Leukemia; Tyrosine Kinase Inhibitor; Withdrawal Syndrome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Substance Withdrawal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples, if not used, will be kept frozen for further exploration if necessary.
  An amendment is produced and approved by ethics commitee in 2021/03/03. It relates to the KIR genes polymorphism and HLA class study in Caen patients in whom NK cell phenotype is available.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with the TKI withdrawal syndrome: There is no intervention. Patients will stop their tyrosine kinase inhibitor yielding to 2 subsets: patients with or without the TKI withdrawal syndrome.
- Group without the TKI withdrawal syndrome: As abovementioned.

SUMMARY:
Patients who suffer from chronic myeloid leukemia are treated by tyrosin kinase inhibitors (TKI) saying imatinib, nilotinib, dasatinib, bosutinib and ponatinib. These drugs are highly efficient with excellent response allowing some patients to definitely stop their cancer treatment. However, in 30% of cases, when the treatment is stopped, pains could arise in shoulders, hips, joints… These symptoms occurring after the withdrawal of a drug are odd and biologically unexplained so far. This study seeks to discover the biological factors behind these symptoms called 'TKI withdrawal syndrome' by the scientific community.

DETAILED DESCRIPTION:
The success of TKI in the treatment of chronic myeloid leukemia is undeniable. Indeed, since the advent of imatinib in 2000 and the subsequent 4 other TKIs, this once fatal disease has become just another chronic disease with patient life expectancy close to the general population. Lifelong TKI therapy offers an 'operational cure' which means quiescent BCR-ABL leukemic stem cells are not eradicated but only controlled.

This statement was challenged in 2008 by the French 'STIM' study in which patients with undetectable BCR-ABL were proposed to discontinue their imatinib: 40% of these patients successfully achieved treatment free remission (TFR) with no recurrence of the disease. These figures are confirmed by the Australian 'TWISTER' study. The resumption of Imatinib therapy was triggered by the positivity of BCR-ABL. In the A-STIM study, the loss of major molecular response is the main criteria to resume imatinib. Accordingly, TFR was a success in 60% of patients. Similar figures was published with second generation TKIs with the same criteria.

In the light of these studies, it is clear that the fields have moved to a more ambitious goal than the operational cure, without the need for remaining on TKI.

Paradoxically, a new syndrome emerged from the Sweden group in 2014: 'the TKI withdrawal syndrome. It consisted of musculoskeletal pains resembling the Polymyalgia Rheumatica in CML patients after discontinuation of Imatinib. It occurred within 6 weeks in 30% of the patients who went on stopping imatinib. Patients with severe pain responded to 10-20 mg of prednisolone. Similar manifestations were described in the European 'EuroSki' study. No explanation was found.

It is well known that TKIs have off-target effects. In addition to BCR-ABL, they inhibit c-Kit, SRC, PDGFR, BTK, TEC, NFKB pathways resulting in anti-inflammatory effects. They can also cause disturbances in electrolyte balance (hypophosphatemia) and bone metabolism. Some research teams have correlated the success of TFR to the increase in cytotoxic NK cells and production IFN and TNFα.

Is the TKI withdrawal syndrome a rebound phenomenon from these off-target effects with excessive release of some cytokines? Of note, an Italian team showed in 4 out of 8 patients with WS an increase of PDGFβ (in 1 patient there was also increase in IL6, TGFβ and VEGF). But no tests were performed in the other patients who stopped TKI and did not presented with the WS as comparison.

Here, the proposed study concerns any CML patient candidate for TKI discontinuation. Will prospectively be checked a number of cytokines and biological factors susceptible to contribute to the clinical features taking into account the off-target effects of TKIs. Therefore, the investigators could compare the variation in a potentially involved cytokine within patients with or without withdrawal syndrome. In addition, the study will prospectively provide a broader description of TKI WS using Brief pain Inventory (BPI) questionnaire.

Eventually, cytokines, inflammatory and bone markers will be dosed at diagnosis and every month during 3 months corresponding to the timeframe in which the withdrawal syndrome is due to occur. A variation of 20% (increase or decrease) in whatever marker(s) will be considered significant if it is (or they are) observed in the group with "TKI withdrawal (TKI WS)" but not in the group without "TKI WS". Pathophysiological explanation of this syndrome could be assumed later taking into account the clinical presentation partly explored by the pain questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Adult CML patient candidate for TKI discontinuation.
* Performans status : 0-2
* Patient provided with information

Exclusion Criteria:

* Patient unable to fulfill the questionnaires
* Patient suffering from demantia
* Patient treated with any cytokine antagonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns patients suffering from Chronic myeloid leukemia treated with TKI (Imatinib, Nilotinib, dasatinib, bosutinib or Ponatinib) for at least 5 years with deep molecular response (MR4) for at least 2 years who agree to stop their drug. Other situation of TKI discontinuation. Five cities are participating in the study: CHU de Caen, CHU d'Amiens, CHU de Clermont-Ferrand, Centre Henri Becquerel de Rouen et le CH de Valenciennes.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Measurement of cytokines: | at diagnosis and every month during 3 months
  Measurement of cytokines: A variation of 20% in a given marker will be significant if it is observed in the group with "TKI WS" but not in the group without "TKI WS". Of note, the patient will be his own witness.
  . In picogram/milliliter (pg/ml): IL2,IL 6, IL10, IL15, TGFβ,TNFα, IFNγ, VEGF, PDGFβ,
Measurement of cytokines: | at diagnosis and every month during 3 months
  In nanogram/milliliter (ng/ml) : Osteoprotegerin
Measurement of cytokines: | at diagnosis and every month during 3 months
  • In microgram/liter (µg/l): Tryptase
Inflammatory markers: | at diagnosis and every month during 3 months
  C reactive protein (milligramme/liter)
Inflammatory markers: | at diagnosis and every month during 3 months
  In international Unit/ liter (IU/l) Rheumatoid factor,
Inflammatory markers: | at diagnosis and every month during 3 months
  In international Unit/ liter (IU/l) Creatinine phosphokinase
bone metabolism markers | at diagnosis and every month during 3 months.
  In microgram/ liter : Cross-laps
bone metabolism markers | at diagnosis and every month during 3 months.
  In microgram/ liter : Procollagen 1
bone metabolism markers | at diagnosis and every month during 3 months.
  PTH (ParaTHormon) (nanogram/Liter)
bone metabolism markers | at diagnosis and every month during 3 months.
  In millimole/Liter: Phosphates
bone metabolism markers | at diagnosis and every month during 3 months.
  In millimole/Liter: Calcium.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) questionnaire | 12 months
  It will help to define the WS thanks to the calculation of the score of pain intensity. The score will be checked at the time the TKI is stopped (baseline) and then every month. Any increase of at least 2 points compared to the baseline will be significant enough to conclude to the TKI WS.
  Pain intensity score is the mean of the scores of the four following questions in which the number 0 confers to "No pain" and 10 to "Pain as bad as the patient can imagine":
  * Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last week.
  * Please rate your pain by marking the box beside the number that best describes your pain at its least in the last week
  * Please rate your pain by marking the box beside the number that best describes your pain on average
  * Please rate your pain by marking the box beside the number that tells how much pain you have right now
QDSA questionnaire | 12 months
  It derives from the McGill questionnaire and describes the type of pain rated by the patient: None = 0; Mild = 1 Moderate =2 Severe = 3. It will complete the BPI questionnaire by giving precision on the type of pain:
  -Throbbing, Shooting, Stabbing, Sharp ...
QLQ C-30 questionnaire | 12 months
  It will explore the quality of life every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyacinthe JOHNSON-ANSAH, Dr, Principal Investigator — UNIVERSITY HOSPITAL of CAEN
Locations (1):
- University hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
Not apllicable

REFERENCES:
- [Background] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Background] Rousselot P, Charbonnier A, Cony-Makhoul P, Agape P, Nicolini FE, Varet B, Gardembas M, Etienne G, Rea D, Roy L, Escoffre-Barbe M, Guerci-Bresler A, Tulliez M, Prost S, Spentchian M, Cayuela JM, Reiffers J, Chomel JC, Turhan A, Guilhot J, Guilhot F, Mahon FX. Loss of major molecular response as a trigger for restarting tyrosine kinase inhibitor therapy in patients with chronic-phase chronic myelogenous leukemia who have stopped imatinib after durable undetectable disease. J Clin Oncol. 2014 Feb 10;32(5):424-30. doi: 10.1200/JCO.2012.48.5797. Epub 2013 Dec 9. PMID 24323036
- [Background] Richter J, Soderlund S, Lubking A, Dreimane A, Lotfi K, Markevarn B, Sjalander A, Saussele S, Olsson-Stromberg U, Stenke L. Musculoskeletal pain in patients with chronic myeloid leukemia after discontinuation of imatinib: a tyrosine kinase inhibitor withdrawal syndrome? J Clin Oncol. 2014 Sep 1;32(25):2821-3. doi: 10.1200/JCO.2014.55.6910. Epub 2014 Jul 28. No abstract available. PMID 25071107
- [Background] Galimberti S, Fontanelli G, Barsotti S, Ricci F, Guerrini F, Barate C. Increased values of the circulating PDGFbeta sustains the "withdrawal syndrome" after tyrosine kinase inhibitor discontinuation in patients affected by chronic myeloid leukemia. Blood Cells Mol Dis. 2015 Oct;55(3):211-2. doi: 10.1016/j.bcmd.2015.06.010. Epub 2015 Jun 23. No abstract available. PMID 26227847